CLINICAL TRIAL: NCT04854018
Title: An Open Label, Single Centre, Single Arm, Prospective Feasibility Study Evaluating the Effectiveness of Near-infrared Fluorescence (NIRF) Using Indo-cyanine Green (ICG) in Minimally Invasive Paediatric Oncology Surgery (MIS)
Brief Title: Indo-cyanine Green (ICG) in Paediatric Oncology MIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20/BC/SME/PO/473
Record Dates: First submitted 2021-02-05; First posted 2021-04-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-04

CONDITIONS: Pediatric Renal Tumor; Metastatic Osteosarcoma; Metastatic Ewing Sarcoma; Pulmonary Metastasis; Rhabdomyosarcoma; Non-Rhabdo. Soft Tissue Sarcoma
Keywords: Indocyanine green; Near Infra-red fluoroscopy; pediatric; oncology; minimal access surgery; Wilms
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Sarcoma; Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: open label, single centre, single arm, prospective feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Injection of Indocyanine Green at doses detailed on summary of product characteristics for each age range
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Intravenous or intraparenchymal injection
  Other Names: Verdye; Diagnostic Green

SUMMARY:
Indo-cyanine green (ICG) is a dye that has been used for a variety of adult and paediatric uses since 1956. Over the past few years, near infrared (NIRF) technology has been developed which allow is use as a fluorescence agent during surgery. It has been used increasingly in the field of adult oncology surgery and has been shown to increase the efficacy of this surgery.

The aim of this study is to evaluate the use of NIRF and ICG during specific minimally invasive surgery (MIS) procedures within paediatric oncology surgery. Their use will complement existing surgical techniques rather than replace them.

Given the published advantages in adults this study aims to provide evidence of feasibility in the paediatric patients with cancer.

DETAILED DESCRIPTION:
The purpose of this study is to show the feasibility of using ICG in combination with NIRF and MIS in paediatric oncology surgery. It has been used increasingly over the past few years for a range of adult oncology surgical indications including tumour margin identification, lymph node identification and pulmonary metastectomy. It will be investigated in three groups of patients in our study:

1. Tumour margin identification-Identifying the margins of a tumour intra-operatively is crucial for many paediatric cancers. Incomplete resections or resections with involved margins often require upstaging of treatment with more intensive chemotherapy or radiotherapy. ICG will be injected intravenously and then NIRF will be used intermittently until fluorescence is achieved and an evaluation of the tumour and its margins will be performed.
2. Lymph node identification - It is standard of care for most oncology resections to remove lymph nodes that are suspected to be involved with tumour. Both SIOP and COG recommend the removal of 7 or more lymph nodes during a nephrectomy for Wilm's tumour although this is often not achieved. IGC will be injected directly into the tumour (or the adjacent tissue in 2-4 places) and then NIRF will be used intermittently until fluorescence is achieved. An evaluation of the tumour and any fluorescent lymph nodes will then take place and any fluorescent lymph nodes will be removed.
3. Pulmonary metastectomy - Many paediatric cancers including Wilm's tumour have a propensity to metastasise to the lungs. Removal of all lung metastases is important as it has the potential to down-stage tumours, obviating the need for pulmonary radiotherapy.

Modern radiology techniques can identify lesions as small as 1mm which are often not palpable at the time of surgery. Relying on finger palpation requires patients to have a thoracotomy with all of the associated complications. ICG will be injected intravenously and then NIRF will be combined with MIS to identify any fluorescent lesions. The location of any lesions will be compared with those seen on pre-surgical imaging (current standard practice).

For all three groups of patients, the use of ICG and NIRF will complement rather than replace existing surgical technique in patients who require surgery already. Data will be collected on the number of lesions which do/do not fluoresce as well as the histology of lesions removed. They will be separated into lesions which do not fluoresce, lesions which were removed before fluorescence (they will be checked for ex-vivo fluorescence) and fluorescing lesions so that the histological characteristics of each group can be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 day and 15 years 365 days
* Have a diagnosis of an intra-abdominal, retroperitoneal or intra-thoracic tumour or pulmonary metastases
* Require surgery as part of their treatment
* Tumour or metastasis suitable for MIS resection based on assessment of the pre-operative imaging

Exclusion Criteria:

* Allergic to ICG
* Allergic to iodine or iodides
* Due to receive radioactive iodine as part of a treatment
* Hyperthyroidism
* Unwilling to participate
* Chronic Kidney Disease stage V

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of fluorescent nodes resected during minimally invasive tumour nephrectomy | Until the end of surgery, 2 hours
  Number of fluorescent nodes resected per patient
Is Fluorescent guided tumour resection easier than non-fluorescent guided. | until the end of surgery, 2 hours
  Subjective surgeon analysis of intra-operative conditions on a Likert scale per patient
To evaluate if NIRF and ICG allow detection of pulmonary metastases | until the end of surgery, 2 hours
  Comparison of number of lesions seen on CT with those seen with fluoroscopy per patient

SECONDARY OUTCOMES:
To evaluate if fluorescent nodes or metastases are more likely to contain viable tumour | until histopathology is reported, 2 weeks
  Number of fluorescent nodes and metastases containing viable tumour per patient

CONTACTS AND LOCATIONS:
Overall Officials: Max Pachl, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (1):
- Birmingham children's hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pachl MJ. Fluorescent Guided Lymph Node Harvest in Laparoscopic Wilms Nephroureterectomy. Urology. 2021 Dec;158:189-192. doi: 10.1016/j.urology.2021.09.015. Epub 2021 Oct 2. PMID 34606881